CLINICAL TRIAL: NCT03779386
Title: Music During Labor and Delivery: Randomized Controlled Trial
Brief Title: Trial of Music During Labor and Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 278/18
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-12

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music during labor and delivery (Experimental): Music during labor and delivery
  Interventions: Other: music
- No music during labor and delivery (No Intervention): No music during labor and delivery

INTERVENTIONS:
Other: music — music during labor and delivery
  Arms: Music during labor and delivery

SUMMARY:
The use of music is widely supported in various areas of medicine: first of all in the psychiatric field as in the treatment of autism in children, obtaining surprising results even on Alzheimer's patients, or the unparalleled effect of music on those suffering from depression. To strengthen the thesis of the usefulness of music in medicine there is what is called PNEI, or the psychoneuroendocrinoimmunology. This discipline consists in the study of mutual interactions between mental activity, behavior, nervous system, endocrine system and immune reactivity. The PNEI itself no longer pays attention to the mind with respect to the body, but using the principles of the empirical epistemology of the scientific method strives to clarify those connections that make the nervous system, mind, immunity and hormonal regulation a unique and complex homeostatic control system of the individual, whose synergism would be able to modify certain biological behaviors, such as the transition from a distress to an eustress. This passage would seem to be of particular obstetric interest going to significantly change the course of labor in terms of pain, anxiety and well-being of women. In fact, many women prefer not to resort to partoanalgesia and famaci for pain control during labor.

A recent Cochrane Review analyzed the effectiveness of music in the control of pain in labor, confirming its role in this sense. However, he concluded that the quality of available evidence varied from low to very low, thus highlighting the need for further studies in this area.

Thus, the present study arises with the rational to satisfy this need for further investigation into the positive effects of music on pain in women in labor.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestations;
* term of phisiological pregnancy
* spontaneous labor
* diagnosis of active phase of labor;
* nulliparous between 37 and 42 gestation weeks with cephalic presentation ;
* maternal age between 18 and 45 years.

Exclusion Criteria:

* multiple gestations;
* preterm labor;
* preterm premature rupture of membranes
* induction to delivery labor;
* Hipertensive disorders;
* fetal abnormalities;
* diabetes mellitus;
* intrauterine growth retardation;
* post-term pregnancy;
* multiple vaginal delivery;
* women with an altered state of consciousness, severely ill, mentally disabled;
* women who are unconscious, severly ill, mentally handicapped;
* women under the age of 18 years or over the age of 45 years.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
pain during the active phase | during the labor
  pain assessed with VAS

SECONDARY OUTCOMES:
anxiety during the active phase, second stage, and postpartum | during the labor
  assessed with VAS
pain during second stage, and during postpartum | during the labor
  pain assessed with VAS
postpartum depression | at the time of delivery
  incidence of postpartum depression
episiotomy and lacerations | at the time of delivery
  incidence of episiotomy and lacerations
analgesia | at the time of delivery
  use of analgesia
labor length | during labor
  length of first stage, and second stage of labor
neonatal outcomes | at the time of delivery until 28days of life
  admission to NICU, neonatal death, a composite of outcomes including NEC, IVH, RDS, BPD, ROP, sepsis, N1CU and death. Multiple measurements (i.e. for composite perinatal outcome) will be aggregated to arrive at one reported value (i.e. incidence of composite perianatal outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buglione A, Saccone G, Mas M, Raffone A, Di Meglio L, di Meglio L, Toscano P, Travaglino A, Zapparella R, Duval M, Zullo F, Locci M. Effect of music on labor and delivery in nulliparous singleton pregnancies: a randomized clinical trial. Arch Gynecol Obstet. 2020 Mar;301(3):693-698. doi: 10.1007/s00404-020-05475-9. Epub 2020 Mar 3. PMID 32125522